CLINICAL TRIAL: NCT03402230
Title: Clinical Study of Avmacol® for Detoxification of Tobacco Carcinogens in Heavy Smokers
Brief Title: Broccoli Sprout/Broccoli Seed Extract Supplement in Decreasing Toxicity in Heavy Smokers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2017-02406; NCI-2017-02406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00031; 1711022046 (Other: University of Arizona Cancer Center - Prevention Research Clinic); UAZ2017-09-02 (Other: DCP); N01CN00031 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2018-01-17; First posted 2018-01-18 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cigarette Smoking-Related Carcinoma; Tobacco-Related Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Avmacol lower dose, Avmacol higher dose) (Experimental): Participants receive lower dose broccoli sprout/broccoli seed extract supplement PO daily for 10-14 days. After 10-14 days, participants receive higher dose broccoli sprout/broccoli seed extract supplement PO daily for 10-14 days.
  Interventions: Drug: Broccoli Sprout/Broccoli Seed Extract Supplement; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm II (Avmacol higher dose, Avmacol lower dose) (Experimental): Participants receive higher dose broccoli sprout/broccoli seed extract supplement PO daily for 10-14 days. After 10-14 days, participants receive lower dose broccoli sprout/broccoli seed extract supplement PO daily for 10-14 days.
  Interventions: Drug: Broccoli Sprout/Broccoli Seed Extract Supplement; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Broccoli Sprout/Broccoli Seed Extract Supplement — Given PO
  Other Names: Avmacol
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized early phase I trial studies how well broccoli sprout/broccoli seed extract supplement works in decreasing toxicity in heavy smokers. Broccoli sprout/broccoli seed extract supplement is a dietary supplement made from broccoli sprout and seed extract powder, and may break down some of the cancer causing substances in tobacco smoke and produce substances that may protect cells from tobacco smoke-induced damage in current smokers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether broccoli sprout/broccoli seed extract supplement (Avmacol) increases the urinary excretion of the mercapturic acid of the tobacco carcinogen, benzene, in healthy volunteers who are current heavy smokers.

SECONDARY OBJECTIVES:

I. To determine whether Avmacol increases the urinary excretion of the mercapturic acids of other tobacco carcinogens, including acrolein and crotonaldehyde.

II. To determine whether Avmacol increases the urinary excretion of the mercapturic acids of tobacco carcinogens, normalized by bio-measurement of tobacco exposure.

III. To determine whether Avmacol upregulates the NRF2 target gene transcripts in the buccal cells of current smokers.

IV. To evaluate for a dose-response relationship between Avmacol and the detoxification of tobacco carcinogens and the expression of NRF2 target gene transcripts.

V. To determine the relationship between systemic study agent exposure and biomarker modulation.

EXPLORATORY OBJECTIVES:

I. To determine whether the GSTM1 and GSTT1 genotypes are important genetic modulators of detoxification of tobacco carcinogens with Avmacol treatment.

II. To bank specimens for future research including evaluation of tobacco gene signatures in buccal and nasal epithelium and buccal cell nuclear morphometry.

OUTLINE: Participants are randomized into 1 of 2 arms.

ARM I: Participants receive lower dose broccoli sprout/broccoli seed extract supplement orally (PO) daily for 10-14 days. After 10-14 days, participants receive higher dose broccoli sprout/broccoli seed extract supplement PO daily for 10-14 days.

ARM II: Participants receive higher dose broccoli sprout/broccoli seed extract supplement PO daily for 10-14 days. After 10-14 days, participants receive lower dose broccoli sprout/broccoli seed extract supplement PO daily for 10-14 days.

After completion of study, participants are followed up at 10-14 days.

ELIGIBILITY:
Inclusion Criteria:

* Current tobacco smokers with >= 20 pack years of self-reported smoking exposure and a current average use of >= 10 cigarettes/day
* Karnofsky performance scale >= 70%
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x ULN
* Creatinine =< ULN
* Fertile subjects must use adequate contraception (abstinence, barrier methods, or birth control pills) prior to study entry and for the duration of study participation; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of invasive cancer within the past 2 years, with the exception of excised and cured non-melanoma skin cancer or carcinoma in situ of the cervix
* Chronic, current or recent (within the past 2 weeks) use of systemic steroid doses equivalent to prednisone > 5 mg daily for continued use > 14 days; use of inhaled steroids, nasal sprays, and topical creams for small body areas is allowed
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Avmacol
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2022-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Bauman, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (2):
- United States (2):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona

RESULTS

PARTICIPANT FLOW:
Groups:
- Avmacol Low Dose First, Then High Dose: Participants received lower dose of Avmacol daily for 10-14 days, followed by 10-14 days of washout, and followed by higher dose of Avmacol daily for 10-14 days.
- Avmacol High Dose First, Then Low Dose: Participants received higher dose of Avmacol daily for 10-14 days, followed by 10-14 days of washout, and followed by lower dose of Avmacol daily for 10-14 days.
Period: Overall Study
Arm/Group | Avmacol Low Dose First, Then High Dose | Avmacol High Dose First, Then Low Dose
Started | 25 | 24
Completed | 25 | 23
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Avmacol: Participants who initiated Avmacol intervention
Arm/Group | Avmacol
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 44
  More than one race | 3
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Excretion of the Mercapturic Acid of Benzene Following 4 Tablets Per Day of Avmacol
Description: Change in the overnight urinary excretion the mercapturic acid of benzene following 4 tablets per day of Avmacol. Data presented as ratio of the geometric mean of overnight urinary excretion the mercapturic acid of benzene between post intervention and baseline.
Time Frame: Baseline up to 14 days post intervention
Measure: Number (95% Confidence Interval); unit: data presented as ratio; no unit
Arm/Group | Avmacol
Number analyzed (Participants) | 48
data presented as ratio; no unit | 1.16 [0.998 to 1.344]

2. Primary Outcome: Change in Urinary Excretion of the Mercapturic Acid of Benzene Following 8 Tablets Per Day of Avmacol
Description: Change in the overnight urinary excretion the mercapturic acid of benzene following 8 tablets per day of Avmacol. Data presented as ratio of the geometric mean of overnight urinary excretion the mercapturic acid of benzene between post intervention and baseline.
Time Frame: Baseline up to 14 days post intervention
Measure: Number (95% Confidence Interval); unit: data presented as ratio; no unit
Arm/Group | Avmacol
Number analyzed (Participants) | 48
data presented as ratio; no unit | 1.19 [1.005 to 1.409]

3. Secondary Outcome: Change in the Urinary Excretion of the Mercapturic Acids of Acrolein and Crotonaldehyde
Description: Change following 4 tablets per day and 8 tablets per day of Avmacol wad determined separately. Data presented as ratio of the geometric mean of overnight urinary excretion of the mercapturic acid of acrolein/crotonaldehyde between post intervention and baseline.
Time Frame: Baseline up to 14 days post intervention
Measure: Number (95% Confidence Interval); unit: data presented as ratio; no unit
Groups:
- Avmacol 4 Tablets: Participants received 4 tablets of the study agent PO daily for 10-14 days.
  Broccoli Sprout/Broccoli Seed Extract Supplement: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Questionnaire Administration: Ancillary studies
- Avmacol 8 Tablets: Participants received 8 tablets of the study agent PO daily for 10-14 days.
  Broccoli Sprout/Broccoli Seed Extract Supplement: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Questionnaire Administration: Ancillary studies
Arm/Group | Avmacol 4 Tablets | Avmacol 8 Tablets
Number analyzed (Participants) | 48 | 48
data presented as ratio; no unit
  Urindary excretion of mercapturic acid of acrolein | 1.11 [0.98 to 1.26] | 1.28 [1.06 to 1.53]
  Urinary excretion of mercapturic acid of crotonaldehyde | 1.05 [0.90 to 1.22] | 1.18 [1.02 to 1.37]

4. Secondary Outcome: Change in the NRF2 Target Gene Transcripts
Description: Change in the expression of NQO1 in the buccal cells after 8 tablets per day of Avmacol. Data presented as ratio of the geometric mean of the gene expression of NQO1 between post intervention and baseline.
Time Frame: Baseline up to 14 days post intervention
Measure: Number (95% Confidence Interval); unit: data presented as ratio; no unit
Groups:
- Avmacol 8 Tablets: Participants received 8 tables of Avmacol
Arm/Group | Avmacol 8 Tablets
Number analyzed (Participants) | 48
data presented as ratio; no unit | 1.00 [0.98 to 1.02]

5. Secondary Outcome: Dose-response Relationship Between Avmacol Dose and Detoxification of Tobacco Carcinogens
Description: Dose-response relationship between the Avmacol dose and the detoxification of tobacco carcinogens. Data presented as ratio of percent change of the overnight urinary excretion of mercapturic acid of benzene/acrolein/crotonaldehyde between the 8 tables and 4 tables dose.
Time Frame: Up to 14 days post intervention
Measure: Number (95% Confidence Interval); unit: data presented as ratio; no unit
Arm/Group | Avmacol
Number analyzed (Participants) | 48
data presented as ratio; no unit
  Mercapturic acid of benzene | 1.01 [0.89 to 1.15]
  Mercapturic acid of acrolein | 1.14 [0.95 to 1.36]
  Mercapturic acid of crotonaldehyde | 1.12 [0.95 to 1.32]

6. Secondary Outcome: Systemic Study Agent Exposure
Description: Change in the total urinary levels of sulforaphane and its glutathione-derived metabolites (i.e., the sum of the molar concentrations of sulforaphane and its glutathione-derived metabolites in urine). Data presented as ratio of the geometric mean of the total urinary levels of sulforaphane and its metabolites between post intervention and baseline.
Time Frame: Up to 14 days post intervention
Measure: Number (95% Confidence Interval); unit: data presented as ratio; no unit
Arm/Group | Avmacol 4 Tablets | Avmacol 8 Tablets
Number analyzed (Participants) | 48 | 48
data presented as ratio; no unit | 467.9 [264.7 to 826.9] | 990.0 [592.2 to 1655.1]

7. Other Pre Specified Outcome: GSTM1 and GSTT1 Genotypes
Description: Change in the urinary excretion of the mercapturic acids of tobacco carcinogens by GSTM1 and GSTT1 genotype. Data presented as ratio of the geometric mean of urinary excretion of mercapturic acid of benzene between post intervention and baseline for each genotype.
Time Frame: Up to 14 days post intervention
Population: The data were presented by genotype. Therefore, the number of participants with a particular genotype is a subset of the overall number of participants analyzed.
Measure: Number (95% Confidence Interval); unit: data presented as ratio; no unit
Arm/Group | Avmacol 4 Tablets | Avmacol 8 Tablets
Number analyzed (Participants) | 48 | 48
data presented as ratio; no unit
  Mercapturic acid of benzene in GSTM1-null participants: number analyzed (Participants) | 23 | 23
  Mercapturic acid of benzene in GSTM1-null participants | 1.23 [0.99 to 1.52] | 1.34 [0.98 to 1.84]
  Mercapturic acid of benzene in GSTM1-positive participants: number analyzed (Participants) | 25 | 25
  Mercapturic acid of benzene in GSTM1-positive participants | 1.10 [0.90 to 1.35] | 1.06 [0.93 to 1.21]
  Mercapturic acid of benzene in GSTT1-null participants: number analyzed (Participants) | 8 | 8
  Mercapturic acid of benzene in GSTT1-null participants | 0.75 [0.54 to 1.04] | 1.16 [0.89 to 1.51]
  Mercapturic acid of benzene in GSTT1-positive participants: number analyzed (Participants) | 40 | 40
  Mercapturic acid of benzene in GSTT1-positive participants | 1.26 [1.08 to 1.47] | 1.20 [0.98 to 1.45]

ADVERSE EVENTS:
Time Frame: Two weeks of agent intervention
Groups:
- High Dose: 8 Tablets of Broccoli Sprout/Broccoli Seed Extract Per Day for 14 days
- Low Dose: 4 Tablets of Broccoli Sprout/Broccoli Seed Extract Per Day for 14 days
Arm/Group | High Dose | Low Dose
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/48
Other Adverse Events (participants affected / at risk) | 26/49 | 14/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=49) | Low Dose (N=48)
Myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=49) | Low Dose (N=48)
Diarrhea (Gastrointestinal disorders) | 10 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 7 | 3
Gastrointestinal disorders, other (Gastrointestinal disorders) | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT03402230/Prot_SAP_000.pdf